CLINICAL TRIAL: NCT01665482
Title: Effects of Dietary Fats on Cardiovascular Health and Insulin Sensitivity in Subjects With Abdominal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PD155/11
Record Dates: First submitted 2012-08-12; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Inflammation; Insulin Sensitivity
Keywords: Inflammation; Insulin sensitivity; Interleukin-6 (IL-6); C-peptide; Saturated fatty acid (SFA); Monounsaturated fatty acid (MUFA); Carbohydrate (CARB)
MeSH Terms: conditions — Inflammation; Insulin Resistance | interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saturated fat rich diet (Active Comparator)
  Interventions: Other: A 2000 kcal test meal
- Monounsaturated fat rich diet (Active Comparator)
  Interventions: Other: A 2000 kcal test meal
- Carbohydrate/ Low fat diet (Active Comparator)
  Interventions: Other: A 2000 kcal test meal which accounts for 7% fat exchange with carbohydrate

INTERVENTIONS:
Other: A 2000 kcal test meal
  Arms: Monounsaturated fat rich diet; Saturated fat rich diet
Other: A 2000 kcal test meal which accounts for 7% fat exchange with carbohydrate
  Arms: Carbohydrate/ Low fat diet

SUMMARY:
Rationale: It is well established that increased intake of saturated fatty acids (SFA) is associated with incidence of cardiovascular heart disease (CHD). This effect is mediated by dietary saturated fat's impact on fasting plasma cholesterol levels. Research is needed to clarify the association between dietary fatty acids and metabolic risk markers beyond lipid profile. World Health Organisation (WHO) has recommended reduced intake of SFA with energy replacement from monounsaturated fatty acids (MUFA) or carbohydrates (CARB). However, limited evidence is available on the effects of dietary fatty acids on insulin sensitivity and secretion. The current study is designed to investigate the effects of SFA versus MUFA versus CARB on insulinemic response and lipid metabolism in healthy individuals with central obesity.

Study design: A randomized, crossover, single blind design study was carried out. The subjects consumed controlled diets for 6 weeks each. They were provided 3 meals per day during weekdays in which SFA, MUFA and CARB diet was assigned to them randomly. Protein content was standardised at 14% energy. The SFA and MUFA diets each provided 31.5% energy intake from fat, with 69% of the total fats replaced by test fats (approximately 49 g/d based on a 2000 kcal basic diet). Each individual fatty acid provided approximately 7% of the total energy intake. The CARB diet provided approximately 34 g/day experimental fat based on a 2000 kcal basic diet. The CARB diet replaced 7 % energy of carbohydrate from total fat with the exchange from oleic acid (C18:1).

Hypothesis: Changing energy from dietary fat (SFA and MUFA) to carbohydrate will influence insulin sensitivity, endothelial and vascular function, pro-inflammatory markers and lipid metabolism differently in individuals with metabolic syndrome. SFA (palm olein) may be comparable with MUFA (high oleic sunflower oil) with regards to its effects on insulin sensitivity, endothelial and vascular function and inflammation

ELIGIBILITY:
Inclusion Criteria:

1. Abdominally obese males and females (waist circumference > 90 cm for male, > 80 cm for female),
2. Age 20-60 years

Exclusion Criteria:

* a medical history of cardiovascular disease, diabetes, dyslipidemia;
* current use of antihypertensive or lipid lowering medication;
* plasma cholesterol > 6.5 mmol/L, TAG > 4.5 mmol/L;
* alcohol intake exceeding a moderate intake (> 28 units per week);
* pregnancy,
* smoker and
* breastfeeding.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 | Baseline, week-5, week-6, week-11, week-12, week-17 and week-18.
C-peptide | Baseline, week-5, week-6, week-11, week-12, week-17 and week-18.

SECONDARY OUTCOMES:
hsCRP | Baseline, week-5, week-6, week-11, week-12, week-17 and week-18.

CONTACTS AND LOCATIONS:
Overall Officials: Teng Kim Tiu, PhD, Principal Investigator — MPOB
Locations (1):
- Malaysia Palm Oil Board (MPOB), Kajang, Selangor, Malaysia

REFERENCES:
- [Derived] Chang LF, Vethakkan SR, Nesaretnam K, Sanders TA, Teng KT. Adverse effects on insulin secretion of replacing saturated fat with refined carbohydrate but not with monounsaturated fat: A randomized controlled trial in centrally obese subjects. J Clin Lipidol. 2016 Nov-Dec;10(6):1431-1441.e1. doi: 10.1016/j.jacl.2016.09.006. Epub 2016 Sep 17. PMID 27919361
- [Derived] Teng KT, Chang LF, Vethakkan SR, Nesaretnam K, Sanders TAB. Effects of exchanging carbohydrate or monounsaturated fat with saturated fat on inflammatory and thrombogenic responses in subjects with abdominal obesity: A randomized controlled trial. Clin Nutr. 2017 Oct;36(5):1250-1258. doi: 10.1016/j.clnu.2016.08.026. Epub 2016 Sep 8. PMID 27642057